CLINICAL TRIAL: NCT06204900
Title: Evaluation Of A Novel Technique To Monitor Neurophysiological Activity During TLIF Surgery Using The Endoscopic Assisted Retropsoas (EARP) Nerve Cuff Electrode and Retractor With A Commercially Available Lumbar Spine Retractor System
Brief Title: A Post-marketing Study to Evaluate a Novel Surgical Monitoring Technique Using the EARP Nerve Cuff in TLIF Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Retropsoas Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EARP-1-1001
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Transforaminal Lumbar Interbody Fusion Surgery
Keywords: TLIF Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Undergoing a single-level or two-level TLIF between L2-S1 (Experimental): During the surgery, the standard monitoring devices and the EARP monitoring study devices and techniques will be used.
  Interventions: Device: Nerve Cuff and Retractor System

INTERVENTIONS:
Device: Nerve Cuff and Retractor System — Endoscopic Assisted Retropsoas (EARP) Nerve Cuff Electrode and an EARP Retractor system to safely monitor lumbar nerve root activity and function during a standard Transforaminal Lumbar Interbody Fusion (TLIF).

SUMMARY:
The purpose of this study is to evaluate the differences (the effectiveness and the safety) between two different nerve and muscle monitoring devices currently available during a TLIF surgery.

The Endoscopic Assisted Retropsoas (EARP) Nerve Cuff Electrode and Retractor surgical and nerve monitoring tools will be used in addition to standard nerve monitoring tools during the surgery. The choice of standard nerve monitoring equipment is based on the decision of the surgeon and technologist and is not dictated by this study.

These tools will be compared with regards to safety and ability to accurately monitor the nervous system during the surgery.

DETAILED DESCRIPTION:
The application of traditional SSEPs and tcMEPs to lumbar nerve root monitoring during TLIF surgery is both challenging and problematic. When applied to lumbar nerve root monitoring, SSEPs and tcMEPs unfortunately suffer in specificity, sensitivity, or both. A surgeon thus cannot confidently rely on these techniques to monitor nerve root function and must guess the likelihood of dysfunction.

Spontaneous EMG (sEMG) is also used to monitor nerve root activity. While sEMG is an excellent indicator of spinal nerve root manipulation, it is a poor diagnostic indicator of dysfunction. 90-95% of sEMG alerts are not associated with dysfunction yielding a high false positive rate and poor specificity, and postoperative deficits are often not associated with sEMG alerts yielding many false negatives and poor sensitivity. The primary utility of sEMG is to use as an indicator of manipulation, which prompts the acquisition of tcMEPs to assess function.

There is a clear need to take the guesswork out of monitoring the functional status of nerve roots at risk during lumbar decompressions and select interbody fusions. During TLIFs, the exiting nerve root is at risk as it courses obliquely across disc space encroaching on the surgical corridor. Standardly, a hand-held retractor is used to retract and protect the nerve root during disc space preparation, implant insertion or even simple decompression. This maneuver and retraction place a particular nerve root at risk, but again, traditional SSEP and tcMEPs are not ideal for monitoring that risk.

The EARP Nerve Cuff Electrode (Retropsoas Technologies) is a novel, Class II, device that is 510(k) cleared by FDA. It conducts electrical signals as a component of intraoperative neuromonitoring, is used with commercially available neuromonitoring systems, and does not stimulate or record the signal itself. The standard connectors at the proximal end interface with the neuromonitoring equipment. The distal nerve cuff electrode partially encircles and contacts the target nerve root. It uses a bipolar configuration to limit current spread. It is available in several inner diameters to accommodate variability in patient nerve root size anatomy.

The EARP Retractor is a Class I device used with a commercially available Retractor system and is only used as an additional 4th blade.

In TLIF surgery, the exiting nerve must be retracted to allow for sufficient access to the intervertebral disc space. The retraction is applied at the medial portion of the nerve root. The application of this retraction may produce activity in the nerve root and/or conduction changes in the nerve root due to temporary manipulation, compression, or ischemia related to the retraction.1

The objective of the study is to demonstrate the ability to safely monitor lumbar nerve root activity and function during retraction using an Endoscopic Assisted Retropsoas (EARP) Nerve Cuff Electrode and an EARP Retractor system during a standard Transforaminal Lumbar Interbody Fusion (TLIF), with improved specificity and sensitivity over traditional monitoring techniques.

ELIGIBILITY:
Inclusion Criteria:

• Undergoing TLIF between L2-S1

Exclusion Criteria:

* Requiring TLIF surgery only at the L5-S1 level
* Acute lumbar spine trauma requiring immediate intervention
* Allergy or contraindication to propofol
* Lower extremity amputation
* Significant lower extremity edema noted on clinical exam
* Current treatment with chemotherapy, radiation, or immunosuppression
* Pregnant, or plans on becoming pregnant in the near future
* History of allergy to titanium, platinum, aluminum, stainless steel, or silicon

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients that experience an Adverse Device Effect (ADE) | From enrollment through the end of the follow-up assessment at week 6
  Adverse device effect (ADE) - Adverse event (AE) judged by the clinician related to the use of an investigational devices. This includes any AE resulting from insufficient or inadequate instructions for use or the deployment, implantation, installation, or operation, or any malfunctioning of the investigational devices and any event resulting from use error or from unintentional misuse of the investigational devices.
Ability of EARP System to alert the surgeon to nerve irritation during surgery compared to standard IONM monitoring techniques | During the TLIF surgery.
  Signal amplitude at baseline, during initial retraction, and maintenance of retraction will be analyzed for changes using a 50% decrease as a surgeon alert. IONM assessments using traditional electrodes: SSEPs, tcMEPs and tfMEP. IONM assessments using EARP cuff: cuff SSEPs, cuff tcMEPs, and cuff tfMEPs.

SECONDARY OUTCOMES:
Evaluate the specificity and sensitivity of alerts to neurological deficits. | From time of surgery through the end of the follow-up assessment at week 6
  Evaluate the sensitivity and specificity of alerts to neurological deficits (by modality and overall). This will include neurological deficits noted on exams as well as a surrogate measure of deficit defined as an alert which resolves with relaxation of retraction.
Assess monitorability of muscles/nerves | During the TLIF surgery.
  Compare the number of evaluable muscles during the surgery by modality and overall.
Assess the change from baseline to end of surgery for each muscle and modality | From enrollment through the end of the follow-up assessment at week 6
  Assess the lower extremity motor deficits post-surgery based on the ipsilateral lower extremity motor exam performed at Baseline, Post-Surgery, and at the 6-week follow-up visit.

OTHER OUTCOMES:
Evaluate the set-up time required for standard IONM monitoring | During the TLIF surgery
  Time for needle placement, tcMEP Baseline acquisition, tfMEP Baseline acquisition, and needle removal will be calculated and compared to set-up of EARP Nerve Cuff
Analyze sEMG activity and any correlations to MEP data and patient-specific characteristics | From enrollment through the end of the follow-up assessment at week 6
  Analyze sEMG activity and any correlations to MEP data and patient-specific characteristics
Characterize retraction, relaxation and release data | During the TLIF surgery
  Characterize retraction, relaxation and release data for the EARP Device
Evaluate total emergence time for anesthetic regimen | During the TLIF surgery
  Evaluate total emergence time for anesthetic regimen

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Poulos, MD, Study Director — Retropsoas Technologies, LLC
Locations (2):
- United States (2):
  - Rothman Orthopaedic Institute, Philadelphia, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  For individual participant data meta-analysis.
  Information can be accessed by contacting the Sponsor directly (contact info TBD)
URL: https://www.inquiry-research.com/